CLINICAL TRIAL: NCT06208956
Title: Effect of Low-dose Dexmedetomidine on Hypotension in Colonoscopy：a Randomized Controlled Trial
Brief Title: A Low Dose Dexmedetomidine in Sedation Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Clinical Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-2105
Record Dates: First submitted 2023-12-11; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. If Ramsay sedation scale score reach 3, colonoscope will be inserted. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg will be administrated as the rescue dose if body movement occur during colonoscopy.
  Interventions: Drug: Dexmedetomidine
- Propofol group (Other): Propofol is administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 until Ramsay score reach 3. During the whole process, propofol is given intermittently to maintain Ramsay score 3 to 4. If body movement happen, propofol 10mg will be administrated every time.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — In the dexmedetomidine group, dexmedetomidine is infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg will be administrated as the rescue dose if body movement occur during colonoscopy.
  Other Names: Dexmedetomidine group
  Arms: Dexmedetomidine group
Drug: Propofol — Propofol is administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 until Ramsay score reach 3. During the whole process, propofol is given intermittently to maintain Ramsay score 3 to 4. If body movement happen, propofol 10mg will be administrated every time.
  Other Names: Propofol group
  Arms: Propofol group

SUMMARY:
104 patients who undergo painless colonoscopy from January 20,2024 to February 29,2024 will be randomized to two groups: propofol group and dexmedetomidine group.

In the dexmedetomidine group,dexmedetomidine is infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. In the propofol group, Propofol is administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1 during the whole process.

DETAILED DESCRIPTION:
104 patients who undergo painless colonoscopy from January 20,2024 to February 29,2024 will be randomized to two groups: propofol group and dexmedetomidine group.

In the dexmedetomidine group,dexmedetomidine is infusion intravenously with a loading dose of 0.5 μg kg-1 for 10 min, then infusion at 0.3 μg kg-1 h-1 according to the ideal body weight of the patient until the end of colonoscopy. In the propofol group, Propofol is administrated 1 mg kg-1 intravenously, then titrated given by 0.5 mg kg-1.For all patients, if Ramsay sedation scale score reach 3, colonoscope will be inserted. During the whole process, maintenance Ramsay score of 3 to 4. Propofol 10 mg will be administrated as the rescue dose if body movement occur during colonoscopy.

The primary outcome is the occurrence of hypotension. Key secondary outcomes are time-weighted average (TWA), area under the threshold (AUT) and cumulative duration of hypotension, as well as the maximum reduction in BP. Other secondary outcomes include(1) the incidence of bradycardia, hypoxemia or body movement；(2) discharge time (from the end of colonoscopy to discharge); (3) patients and endoscopists' satisfaction score (using an 11-point Likert scale, with 0 indicating "very dissatisfied" and 10 indicating "very satisfied"); (4) the incidence of dizziness, fatigue, or nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged above 18 years
2. American Society of Anesthesiologists (ASA) physical status of 1-2
3. Patients scheduled for sedation colonoscopy

Exclusion Criteria:

1. Emergency patients
2. Body weight < 40 kg or >100 kg
3. Allergy to dexmedetomidine, propofol in this trail, a previous adverse reaction to dexmedetomidine or propofol
4. Pregnancy or lactation
5. Drug abusers
6. Participation in other clinical studies within the previous 3 months
7. renal impairment (glomerular filtration rate < 60 ml/min), significant hepatic impairment (ascites, cirrhosis, or with international normalized ratio(INR) >1.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the incidence of hypotension | The time during colonoscopy, an average of 15 minutes
  Hypotension is defined as 20% decrease from baseline systolic blood pressure (SBP) or diastolic blood pressure (DBP), or SBP < 90, and/or DBP < 50 mmHg

SECONDARY OUTCOMES:
Area under the threshold (AUT) of hypotension | The time during colonoscopy, an average of 15 minutes
  AUT=depth of hypotension below (a 20% decrease in baseline SBP or DBP) or (90 mm Hg of SBP or 50 mm Hg of DBP)× time in minutes spent of hypotension. As an example, a patient undergoes colonoscopy that lasts 15 min, in which he experiences 2 episodes of hypotension, all lasting for 1 min and all with a minimal SBP of 80 mm Hg. The AUT = 2 min × (90 -80= 10 mm Hg under the SBP threshold of 90 mm Hg) = 2×10 = 20 mm Hg per minute.
Time-weighted average (TWA) | The time during colonoscopy, an average of 15 minutes
  TWA is calculated as the AUT divided by the total duration of colonoscopy
Cumulative duration of hypotension | The time during colonoscopy, an average of 15 minutes
  The total time of patients experience hypotenion（hpotension defined as 20% decrease from baseline systolic blood pressure (SBP) or diastolic blood pressure (DBP), or SBP < 90, and/or DBP < 50 mmHg)
Maximum reduction in blood pressure (BP) | The time during colonoscopy, an average of 15 minutes
  Maximum reduction in systolic blood pressure (SBP) ,diastolic blood pressure (DBP) and mean arterial pressure (MAP) from baseline
The incidence of bradycardia | The time during colonoscopy, an average of 15 minutes
  Bradycardia is defined as heat rate(HR) <50 beats/min
The incidence of hypoxemia | The time during colonoscopy, an average of 15 minutes
  Hypoxemia is defined as oxygen saturation (SpO2)<90%
The body movement | The time during colonoscopy, an average of 15 minutes
  The twisting of the patient's body due to the stimulation of the colonoscopy, making it difficult to proceed with the procedure
Discharge time | From the end of colonoscopy to discharge，an average of 40 minutes
  From the end of colonoscopy to discharge
Patients satisfaction score | When the patient is fully awake after colonoscopy，an average of 5 minutes
  Using an 11-point Likert scale, with 0 indicating "very dissatisfied" and 10 indicating "very satisfied"
Endoscopists'satisfaction score | At the end of colonoscopy,an average of 15 minutes
  Using an 11-point Likert scale, with 0 indicating "very dissatisfied" and 10 indicating "very satisfied"
The incidence of dizziness | From the end of colonoscopy to discharge，an average of 40 minutes
  The investigators consider it dizziness if patients fell any dizziness
The incidence of fatigue | From the end of colonoscopy to discharge，an average of 40 minutes
  The investigators consider it fatigue if patients fell any fatigue
The incidence of nausea and vomiting | From the end of colonoscopy to discharge，an average of 40 minutes
  The investigators consider it nausea and vomiting if patients fell any nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhou, Study Chair — China, Sichuan West China Hospital

IPD SHARING:
Plan to Share IPD: No